CLINICAL TRIAL: NCT02088177
Title: Open-Label Pilot Study of Long-Acting Injectable Naltrexone Treatment for Cannabis Dependence
Brief Title: Study of Long-Acting Injectable Naltrexone to Treat Cannabis Dependence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6799; DA009236 (Other Grant/Funding Number: National Institutes on Drug Abuse)
Record Dates: First submitted 2014-02-25; First posted 2014-03-14 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Cannabis Dependence
Keywords: Cannabis; Cannabis Dependence; Cannabis Use Disorder; Marijuana; Naltrexone; Long Acting Injectable Naltrexone; Treatment
MeSH Terms: conditions — Marijuana Abuse | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Long-acting injectable naltrexone (Experimental): Two doses of long-acting injectable naltrexone, 380 mg by intramuscular injection in the gluteal muscle at study day 1 and again between study days 28-30.
  Interventions: Drug: Long-acting injectable naltrexone

INTERVENTIONS:
Drug: Long-acting injectable naltrexone — Vivitrol is a long-acting opioid antagonist which blocks opioid agonists from binding at opioid receptors. It be administered as described above.
  Other Names: Vivitrol

SUMMARY:
This is an 8 week, outpatient research study testing the use of long-acting naltrexone (Vivitrol) as a treatment for marijuana dependence. Vivitrol is a medication that is effective in treating dependence on opiates and opioids, and in treating dependence on alcohol. It is FDA approved for these disorders. It is a long-acting medication that contains enough medicine in each injection to last for one month. One way it works is by blocking the effects of opiates, including opiates released by the body in response to drugs and alcohol. In this study, we are interested in testing the effects of Vivitrol in people with marijuana dependence.

Individuals participating in this study will receive two Vivitrol injections, each given four weeks apart, (week 1 and week 5). The injection is given in the muscle of the buttock on one side. Participants will attend clinic visits two times a week during this 8-week study for medical management for drug use and for monitoring of physical and psychological health.

DETAILED DESCRIPTION:
This is an 8 week, outpatient, open-label clinical trial of long-acting injectable naltrexone as a treatment for cannabis dependence.

The purpose of the study will be to evaluate marijuana use patterns and tolerability of long-acting naltrexone in 7 treatment-seeking, cannabis-dependent outpatients; also to assess feasibility of conducting a larger trial with this medication. Cannabis dependent patients will have twice weekly clinic visits where they will receive injections of Vivitrol four weeks apart, in Week 1 and in Week 5. The psychosocial intervention for this study will be Medical Management, designed to facilitate adherence to the study medication and monitoring procedures, as well as to support the participant in achieving his or her marijuana use goals.

Participants will self-report cannabis use, will provide urine toxicology for quantitative assessment of THC (Tetrahydrocannabinol, the active ingredient in marijuana), and will provide serum samples for safety monitoring, and will answer questionnaires and will report on their physical and psychological health weekly.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 - 60 years
* Meets DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, edition IV-TR) criteria for cannabis dependence
* Seeking treatment for cannabis dependence
* Reports using cannabis an average of 5 days per week over the past 28 days
* Capable of giving informed consent and complying with study procedures

Exclusion Criteria:

* Lifetime history of DSM-IV diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder
* Currently meeting DSM-IV criteria for a psychiatric disorder that, according to the investigator's judgment, may require pharmacological or non-pharmacological intervention during the course of the study
* Receiving opioid analgesic medication
* Known history of allergy, intolerance, or hypersensitivity to naltrexone
* Pregnancy, lactation, or failure to use adequate contraceptive methods in female participants who are actively engaging in sexual activity with men
* Unstable medical conditions, such as poorly controlled hypertension or liver disease, which might make participation hazardous
* Chronic pain conditions
* Liver dysfunction as indicated by elevated liver transaminases greater than 2 times the upper limit of normal
* Current DSM-IV diagnosis of substance dependence other than nicotine or cannabis dependence
* Legally mandated to participate in a substance use disorder treatment program
* Risk for suicide

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Notzon, M.D., Principal Investigator — Columbia and NY Psychiatric Institute
Locations (2):
- United States (2):
  - STARS Downtown, Columbia-Presbyterian and New York State Psychiatric Institute, New York, New York
  - STARS clinic, Columbia-New York Presbyterian and New York State Psychiatric Institute, New York, New York

REFERENCES:
- [Result] Johnson BA, Ait-Daoud N, Roache JD. The COMBINE SAFTEE: a structured instrument for collecting adverse events adapted for clinical studies in the alcoholism field. J Stud Alcohol Suppl. 2005 Jul;(15):157-67; discussion 140. doi: 10.15288/jsas.2005.s15.157. PMID 16223067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at the Substance Treatment and Research Service (STARS), a research clinic at Columbia University Medical Center and the New York State Psychiatric Institute in New York, NY. Participant recruitment began in October 2014 and concluded in January 2016, with data collection completed in March 2016.
Pre-assignment Details: All participants were assigned to treatment with injectable naltrexone under open-label conditions. The first injection was given on study day 1.
Groups:
- Open Label Group: open label group receiving injections of long acting naltrexone
Period: Overall Study
Arm/Group | Open Label Group
Started | 12
Completed | 9
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Group
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.42 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 2
  More than one race | 0
  Unknown or Not Reported | 3
education level [Count of Participants; unit: Participants]
  High School | 6
  Some College | 1
  post high school technical training | 1
  College Graduate | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Marijuana Use
Description: Change in marijuana use, as measured by comparing the mean number of self reported days of marijuana use per week in the final study week, which will be week 8 or earlier if the participant discontinues as compared to the mean number of self reported days of marijuana use in week 1
Time Frame: Weeks 1 - 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Open Label Group
Number analyzed (Participants) | 12
days | -1.7 (.51)

2. Primary Outcome: Number of Participants Receiving the Second Injection of Study Medication
Description: The number of participants who accept the second injection at week 5 will be used as one measure of tolerability.
Time Frame: Weeks 1 - 5
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Group
Number analyzed (Participants) | 12
Participants | 6

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Open Label Group
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Group (N=12)
insomnia (General disorders) | 6 (6)
nausea (Gastrointestinal disorders) | 6 (6)
appetite change (Gastrointestinal disorders) | 4 (4)
induration (Injury, poisoning and procedural complications) | 4 (4)
anxiety (Psychiatric disorders) | 3 (3)
vomitting (Gastrointestinal disorders) | 2 (2)
irritability (General disorders) | 2 (2)
fatigue (General disorders) | 1 (1)
headache (General disorders) | 1 (1)
muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
vivid dreams (General disorders) | 1 (1)
diaphoresis (Skin and subcutaneous tissue disorders) | 1 (1)
lightheadedness (General disorders) | 1 (1)
chills (General disorders) | 1 (1)
dry heaves (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Our study is open-label, uncontrolled and with a small sample size, and is not designed to test a priori hypotheses as to the safety, efficacy or effectiveness of our treatment intervention beyond its feasibility for further study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes